CLINICAL TRIAL: NCT05350865
Title: Prevalence, Risk Factor and Clinical Significance of Hepatitis D Virus Infection Among Targeted High Risk Population in Thailand: Nationwide Survey 2022-2024
Brief Title: Thailand HDV Cohort
Status: Recruiting | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other); Thai Red Cross AIDS Research Centre (Other); Siriraj Hospital (Other); Taksin Hospital (Unknown); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 304
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: HDV
Keywords: HBV; HDV; cirrhosis; Thailand
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The participants will have blood test for antiHD, HDV RNA, HBsAg, HBeAg, HBV DNA, antiHCV, and HIV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HDV cohort: Chronic Hepatitis B (HBsAg+) with cirrhosis (APRI >1.5, FIB-4 > 3.25, Fibroscan > 12.5, imaging), PWID with HBV, HIV/HBV, HBV/HCV, aged 18 years and older

SUMMARY:
There is very limited data of HDV in Thailand. As both HDV and HIV can accelerate the HBV course and increased the risk of death, particularly, among those with low CD4 cells/count, therefore, HDV burden in this special population is unmet need. Therefore, this study plans to perform a nationwide survey of the prevalence and predictor of HDV among people uses drugs (PWID) with and without HIV, HBV/HIV (MSM vs non MSM), HBV related cirrhosis. Findinds from this study will provide the scientific community to understand how important HDV is among HBV patients, this could be used to develop strategies for HDV screening and treatment

DETAILED DESCRIPTION:
The prevalence of HDV remains ill-defined, mainly for lack of appropriate testing and screening. As both HDV and HIV can accelerate the HBV course and increased the risk of death, particularly, among those with low CD4 cells/count, therefore, HDV burden in this special population is unmet need. This data will inform the guideline whether HDV screening among HBV/HIV is required. This study has plans to perform a nationwide survey of the prevalence and predictor of HDV among people uses drugs (PWID) with and without HIV, HBV/HIV (MSM vs non MSM), HBV related cirrhosis. This Nationwide survey of HDV is collaboration between Thai liver society, Thai AIDS society, Thai Red Cross AIDS research centre, Faculty of Medicine Chulalongkorn University, and AIDS TB and STI Control Division, Department of Disease control, MOPH Thailand. All findings will be shared and discussed to develop the National guideline for screening, treatment and care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years and older
2. Chronically-infected with HBV, as defined by:

   Positive Hepatitis B surface antigen HBsAg) or HBV DNA result with a subsequent positive HBsAg or HBV DNA result at least 6 months after first positive result
3. Provide signed and dated informed consent form.

Exclusion Criteria:

Non chronic HBV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronically-infected with HBV, as defined by: Positive Hepatitis B surface antigen HBsAg) or HBV DNA result with a subsequent positive HBsAg or HBV DNA result at least 6 months after first positive result
Sampling Method: Non-Probability Sample
Enrollment: 3152 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of HDV | 1 year
  prevalence of HDV in patients with cirrhosis
prevalence of HDV | 1 year
  prevalence of HDV in patients with non cirrhosis
prevalence of HDV | 1 year
  prevalence of HDV in HIV positive people with injecting drug use
prevalence of HDV | 1 year
  prevalence of HDV in HIV negative people with injecting drug use
prevalence of HDV | 1 year
  prevalence of HDV among HBV/HIV men who have sex with men
prevalence of HDV | 1 year
  prevalence of HDV among HBV/HIV cisgender male patients
prevalence of HDV | 1 year
  prevalence of HDV among prisoners
proportion of participants with detectable HDV RNA among seropositive anti HDV | 1 year
  proportion of participants with detectable HDV RNA among seropositive anti HDV with cirrhosis
proportion of participants with detectable HDV RNA among seropositive anti HDV | 1 year
  proportion of participants with detectable HDV RNA among seropositive anti HDV without cirrhosis
proportion of participants with detectable HDV RNA among seropositive anti HDV | 1 year
  proportion of participants with detectable HDV RNA among seropositive anti HDV in PWID with HIV
proportion of participants with detectable HDV RNA among seropositive anti HDV | 1 year
  proportion of participants with detectable HDV RNA among seropositive anti HDV in PWID without HIV
proportion of participants with detectable HDV RNA among seropositive anti HDV | 1 year
  proportion of participants with detectable HDV RNA among seropositive anti HDV with HIV/HBV MSM
proportion of participants with detectable HDV RNA among seropositive anti HDV | 1 year
  proportion of participants with detectable HDV RNA among seropositive anti HDV in HIV/HBV cisgender males
proportion of participants with detectable HDV RNA among seropositive anti HDV | 1 year
  proportion of participants with detectable HDV RNA among seropositive anti HDV in prisoners
predictive risk of HDV infection | 1 year
  predictive risk of HDV infection
HDV subtype | 1 year
  HDV subtype among people with cirrhosis
HDV subtype | 1 year
  HDV subtype among people without cirrhosis
HDV subtype | 1 year
  HDV subtype in PWID with HIV
HDV subtype | 1 year
  HDV subtype in PWID without HIV
HDV subtype | 1 year
  HDV subtype in HBV/HIV MSM
HDV subtype | 1 year
  HDV subtype in HBV/HIV cisgender males
HDV subtype | 1 year
  HDV subtype in prisoners
performance of antiHDV commercial kits | 1 year
  performance of antiHDV commercial kits
prevalence of HDV among HBV/HIV before combination antiretroviral therapy | 1 year
  prevalence of HDV among HBV/HIV before combination antiretroviral therapy
prevalence of HDV among HBV/HIV after combination antiretroviral therapy | 1 year
  prevalence of HDV among HBV/HIV after combination antiretroviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre; Pisit Tangkijvanich, MD, Principal Investigator — Biochemistry, Faculty of Medicine, Chulalongkorn University
Locations (4):
- Thailand (4):
  - HIV-NAT, Thai Red Cross - AIDS Research Centre, Bangkok, Bangkok
  - King memorial Chulalongkorn hospital, Bangkok, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok, Bangkok
  - Taksin Hospital, Bangkok, Bangkok